CLINICAL TRIAL: NCT03392337
Title: An Open-Label, Pilot Study to Evaluate the Efficacy of Narrowband Ultraviolet-B Phototherapy Three Times Weekly for Twelve Weeks in Moderate-to-Severe Psoriasis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC02
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label Narrowband UVB phototherapy (Experimental): Open Label Narrowband UVB phototherapy for 12 weeks.
  Interventions: Device: Narrowband UVB phototherapy

INTERVENTIONS:
Device: Narrowband UVB phototherapy — Ultraviolet B phototherapy

SUMMARY:
A single center study of 30 patient receiving Narrowband UVB phototherapy three times weekly for 12 weeks. Patients will be evaluated through week 36 to evaluate maintenance of response.

DETAILED DESCRIPTION:
30 subjects will be treated with increasing doses of Narrowband Ultraviolet phototherapy three times weekly for 12 weeks. Patients will then be evaluated every 6 weeks through week 36 to determine maintenance of response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥ 18 years of age.
2. Diagnosis of chronic plaque-type psoriasis for at least 6 months
3. Moderate to Severe plaque psoriasis as defined by BSA ≥10 PASI ≥12 IGA ≥3
4. Able to give written informed consent prior to performance of any study related procedures
5. Subject is able to attend Narrowband UVB phototherapy sessions three times a week and all other protocol specified visits
6. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic, and/or guttate psoriasis) or drug induced psoriasis
2. History of photosensitivity
3. Subject has used ustekinumab and/or anti-IL-17 biologic therapy within 24 weeks or other experimental or commercially available biologic immune modulator(s) within 12 weeks prior to the first IP dose.
4. Use of any investigational drug within 4 weeks prior to randomization, or within 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
5. Use of oral systemic medications for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin, apremilast and cyclosporine).
6. Patient used topical therapies to treat within 2 weeks of the Baseline Visit (includes, but not limited to, topical corticosteroids, vitamin D analogs, or retinoids).
7. Initiated within 3 months, planned initiation of, or changes to, concomitant medications that could affect psoriasis vulgaris (e.g. beta blockers, antimalarial drugs, lithium, ACE inhibitors ) during the trial
8. Active infections requiring antibiotics in the 2 weeks prior to Baseline
9. Patient received UVB phototherapy within 4 weeks of Baseline.
10. Patient received PUVA phototherapy within 4 weeks of Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area severity index score | 12 weeks
  PASI 75

SECONDARY OUTCOMES:
Physicians Global Assessment | 12 weeks
  PGA improvement
Body Surface Area | 12 weeks
  BSA improvement
Physician's Global Assessments multiplied by Body surface area | 12 weeks
  PGA x BSA

CONTACTS AND LOCATIONS:
Locations (1):
- Elise Nelson, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No